CLINICAL TRIAL: NCT05053425
Title: Clinical Study of Bcl-2 Inhibitors Combined With Azacytidine and Chemotherapy in Elderly Patients With Previously Untreated Acute Myeloid Leukemia
Brief Title: Bcl-2 Inhibitors Combined With Azacytidine and Chemotherapy in Elderly Patients With Previously Untreated AML
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: LanZhou University (Other)
Responsible Party: Principal Investigator, Long Zhao, Doctor-in-charge, Master of Medicine, LanZhou University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSBCL2; ChiCTR2100045330 (Registry Identifier: Chinese Clinical Trial Registry)
Record Dates: First submitted 2021-09-16; First posted 2021-09-22 (Actual); Last update posted 2022-04-26 (Actual); Status verified 2022-04

CONDITIONS: Acute Myeloid Leukemia
Keywords: Acute Myeloid Leukemia; Bcl-2 Inhibitors; Azacytidine; Chemotherapy
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — venetoclax; Azacitidine; Cladribine; Cytarabine; Idarubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Venetoclax group (Experimental): Induction therapy: venetoclax d1 100mg, d2 200mg, d3-28 400mg, po; azacytidine 75mg/m2, d1-7, sc.
  Consolidation therapy: Regimen A or B was chosen according to the wishes of the patients. In addition, venetoclax was used for 14 days for positive minimal residual disease(MRD) and 7 days for MRD negative.
  regimen A: the first two cycles: venetoclax 400mg, d1-7/14, po; cladribine 5mg/m2, d1-3, ivgtt; cytarabine 10mg/m2, q12h, d1-10, sc; the last two cycles: venetoclax 400mg, d1-7/14, po; cytarabine 0.5-1.0g/m2, d1-3, ivgtt; regimen B: the first two cycles: venetoclax 400mg, d1-7/14, po; cytarabine 100mg/m2, d1-5/7, ivgtt; idarubicin 8mg/m2, d1-2/3, ivgtt; the last two cycles: venetoclax 400mg, d1-7/14, po; cytarabine 0.5-1.0g/m2, d1-3, ivgtt; If the patient's ECOG performance status ≥2,the reduction of regimen IA(cytarabine+idarubicin)was 5+2.
  Maintenance therapy: azacytidine 75mg/m2, d1-7, sc.
  Interventions: Drug: Venetoclax; Drug: Azacitidine; Drug: Cladribine; Drug: Cytarabine; Drug: Idarubicin

INTERVENTIONS:
Drug: Venetoclax — given po.
  Other Names: ABT-199
Drug: Azacitidine — given sc.
  Other Names: 5-Azacytidine
Drug: Cladribine — given ivgtt.
  Other Names: 2-CdA
Drug: Cytarabine — given sc or ivgtt.
  Other Names: Ara-c
Drug: Idarubicin — given ivgtt.
  Other Names: Idamycin®

SUMMARY:
In this prospective study, 30 newly untreated elderly patients with acute myeloid leukemia(AML) who were not suitable for standard chemotherapy were enrolled to observe the efficacy and side effects of venetoclax (VEN) combined with azacytidine (AZA) and chemotherapy in newly treated elderly patients with AML. Overall survival (OS), complete remission rate/complete remission with incomplete recovery of blood cell count (CR/ CRi) were used as the primary endpoints, and time to response (TTR), duration of response (DOR), mortality, and recurrence rate were used as secondary endpoints,and the incidence of adverse events were evaluated.

DETAILED DESCRIPTION:
Induction therapy: venetoclax d1 100mg, d2 200mg, d3-28 400mg, po; azacytidine 75mg/m2, d1-7, sc. Consolidation therapy: Regimen A or B was chosen according to the wishes of the patients. In addition, venetoclax was used for 14 days for positive minimal residual disease(MRD) and 7 days for MRD negative.

regimen A: the first two cycles: venetoclax 400mg, d1-7/14, po; cladribine 5mg/m2, d1-3, ivgtt; cytarabine 10mg/m2, q12h, d1-10, sc; the last two cycles: venetoclax 400mg, d1-7/14, po; cytarabine 0.5-1.0g/m2, d1-3, ivgtt; regimen B: the first two cycles: venetoclax 400mg, d1-7/14, po; cytarabine 100mg/m2, d1-5/7, ivgtt; idarubicin 8mg/m2, d1-2/3, ivgtt; the last two cycles: venetoclax 400mg, d1-7/14, po; cytarabine 0.5-1.0g/m2, d1-3, ivgtt; If the patient's ECOG performance status ≥2, the reduction of regimen IA(cytarabine+idarubicin)was 5+2. Maintenance therapy: azacytidine 75mg/m2, d1-7, sc.

ELIGIBILITY:
Inclusion Criteria:

1. The elderly patients(≥ 60) with AML diagnosed according to WHO criteria;
2. Participants are ineligible for induction regimen;
3. The Eastern Cooperative Oncology Group (ECOG) performance status is 0-3;
4. The patients and their families agree and sign the informed consent form.

Exclusion Criteria:

1. Previous treatment for AML (including hypomethylating agents and other chemotherapy drugs);
2. Infiltration of the central nervous system;
3. Drugs use history affecting CYP3A within 7 days before enrollment;
4. participants considered by the investigator to be unsuitable for inclusion.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-10-20 (Actual); Primary Completion 2023-01-18 (Estimated); Study Completion 2023-03-18 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | up to 16 months.
  Overall survival will be defined as the number of days from the date of first dose to the date of death.
CR/CRi | up to 16 months.
  To assess the percentage of patients achieving CR/CRi according to the International Working Group criteria for AML.

SECONDARY OUTCOMES:
Time to response | up to 16 months.
  To assess the percentage of patients achieving CR/CRi or partial remission (PR) according to the International Working Group criteria for AML.
Duration of response | up to 16 months.
  Duration of response will be defined as the number of days from the date of first response per the IWG criteria for AML to the earliest recurrence or progressive disease.
Mortality | up to 16 months.
  The proportion of patients from enrollment to death was recorded.
Recurrence rate | up to 16 months.
  Record the proportion of patients with recurrence in the study.
Adverse events | Adverse events were assessed weekly during the first and second cycles, and every two cycles thereafter (each cycle is 28 days), up to 16 months.
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Long Zhao, M.M., Principal Investigator — The First Hospital of Lanzhou University,Lanzhou,Gansu,China
Locations (1):
- Long Zhao, Lanzhou, Gansu, China

IPD SHARING:
Plan to Share IPD: No